CLINICAL TRIAL: NCT00523341
Title: An Open Label, Single Arm, Extension Study to Evaluate the Long Term Safety and Sustained Efficacy of Denosumab (AMG162) in the Treatment of Postmenopausal Osteoporosis
Brief Title: Extension Study to Evaluate the Long Term Safety and Efficacy of Denosumab in the Treatment of Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060289
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Results first posted 2016-07-12 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Osteopenia; Osteoporosis
Keywords: postmenopausal osteoporosis; low bone density; fractures; low bone mass
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Osteoporosis, Postmenopausal; Fractures, Bone | interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Denosumab (Experimental): Participants received a 60 mg subcutaneous injection of denosumab every 6 months for seven years.
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: Denosumab — Administered by subcutaneous injection once every 6 months.
  Other Names: AMG 162; Prolia

SUMMARY:
The primary objective was to describe the safety and tolerability of up to 10 years or 7 years denosumab administration as measured by adverse event monitoring, immunogenicity and safety laboratory parameters in participants who previously received denosumab or placebo, respectively.

ELIGIBILITY:
Postmenopausal women who have attended the 20030216 (NCT00089791) study month 36 visit will be eligible to participate if they meet the inclusion and exclusion criteria given below.

Inclusion Criteria

* Subjects must sign the informed consent before any study specific procedures are performed and agree to receive denosumab 60 mg subcutaneous injection every 6 months
* Subjects must not have discontinued investigational product during the 20030216 study and must have attended the 20030216 study month 36 visit
* Subjects must be re-consented prior to (or at) the 24 month visit for participation beyond month 24.

Exclusion Criteria

* Permanently non-ambulatory subjects (use of an assistive device eg, cane, walker, etc. is permitted)
* Missed 2 or more investigational product doses during the 20030216 study
* Any disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or comply with study procedures
* Developed sensitivity to mammalian cell derived drug products during the 20030216 study
* Unable to tolerate calcium supplementation during the last 6 months of participation in the 20030216 study (between the month 30 and month 36 20030216 study visits)
* Currently receiving any investigational product other than denosumab or having received any investigational product during the 20030216 study
* Current use of the following osteoporosis agents: bisphosphonates, calcitonin, fluoride, parathyroid hormone, selective estrogen receptor modulators, systemic oral or transdermal estrogen (except vaginal preparations and estrogen creams which are acceptable), strontium, or tibolone
* For bone biopsy sub-study subjects only: known or suspected sensitivity or contraindication to tetracycline derivatives

Ages: 60 Years to 94 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4550 (Actual)
Dates: Start 2007-08-07 (Actual); Primary Completion 2015-07-19 (Actual); Study Completion 2015-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Cummings SR, Ferrari S, Eastell R, Gilchrist N, Jensen JB, McClung M, Roux C, Torring O, Valter I, Wang AT, Brown JP. Vertebral Fractures After Discontinuation of Denosumab: A Post Hoc Analysis of the Randomized Placebo-Controlled FREEDOM Trial and Its Extension. J Bone Miner Res. 2018 Feb;33(2):190-198. doi: 10.1002/jbmr.3337. Epub 2017 Nov 22. PMID 29105841
- [Background] Dempster DW, Brown JP, Fahrleitner-Pammer A, Kendler D, Rizzo S, Valter I, Wagman RB, Yin X, Yue SV, Boivin G. Effects of Long-Term Denosumab on Bone Histomorphometry and Mineralization in Women With Postmenopausal Osteoporosis. J Clin Endocrinol Metab. 2018 Jul 1;103(7):2498-2509. doi: 10.1210/jc.2017-02669. PMID 29672714
- [Background] Bone HG, Wagman RB, Brandi ML, Brown JP, Chapurlat R, Cummings SR, Czerwinski E, Fahrleitner-Pammer A, Kendler DL, Lippuner K, Reginster JY, Roux C, Malouf J, Bradley MN, Daizadeh NS, Wang A, Dakin P, Pannacciulli N, Dempster DW, Papapoulos S. 10 years of denosumab treatment in postmenopausal women with osteoporosis: results from the phase 3 randomised FREEDOM trial and open-label extension. Lancet Diabetes Endocrinol. 2017 Jul;5(7):513-523. doi: 10.1016/S2213-8587(17)30138-9. Epub 2017 May 22. PMID 28546097
- [Background] Ferrari S, Eastell R, Napoli N, Schwartz A, Hofbauer LC, Chines A, Wang A, Pannacciulli N, Cummings SR. Denosumab in postmenopausal women with osteoporosis and diabetes: Subgroup analysis of FREEDOM and FREEDOM extension. Bone. 2020 May;134:115268. doi: 10.1016/j.bone.2020.115268. Epub 2020 Feb 10. PMID 32058020
- [Background] Ferrari S, Lewiecki EM, Butler PW, Kendler DL, Napoli N, Huang S, Crittenden DB, Pannacciulli N, Siris E, Binkley N. Favorable skeletal benefit/risk of long-term denosumab therapy: A virtual-twin analysis of fractures prevented relative to skeletal safety events observed. Bone. 2020 May;134:115287. doi: 10.1016/j.bone.2020.115287. Epub 2020 Feb 21. PMID 32092479
- [Background] Kendler DL, Chines A, Brandi ML, Papapoulos S, Lewiecki EM, Reginster JY, Munoz Torres M, Wang A, Bone HG. The risk of subsequent osteoporotic fractures is decreased in subjects experiencing fracture while on denosumab: results from the FREEDOM and FREEDOM Extension studies. Osteoporos Int. 2019 Jan;30(1):71-78. doi: 10.1007/s00198-018-4687-2. Epub 2018 Sep 22. PMID 30244369
- [Background] Watts NB, Brown JP, Papapoulos S, Lewiecki EM, Kendler DL, Dakin P, Wagman RB, Wang A, Daizadeh NS, Smith S, Bone HG. Safety Observations With 3 Years of Denosumab Exposure: Comparison Between Subjects Who Received Denosumab During the Randomized FREEDOM Trial and Subjects Who Crossed Over to Denosumab During the FREEDOM Extension. J Bone Miner Res. 2017 Jul;32(7):1481-1485. doi: 10.1002/jbmr.3119. Epub 2017 Apr 3. PMID 28277603
- [Background] Watts NB, Grbic JT, Binkley N, Papapoulos S, Butler PW, Yin X, Tierney A, Wagman RB, McClung M. Invasive Oral Procedures and Events in Postmenopausal Women With Osteoporosis Treated With Denosumab for Up to 10 Years. J Clin Endocrinol Metab. 2019 Jun 1;104(6):2443-2452. doi: 10.1210/jc.2018-01965. PMID 30759221
- [Background] Adachi JD, Bone HG, Daizadeh NS, Dakin P, Papapoulos S, Hadji P, Recknor C, Bolognese MA, Wang A, Lin CJF, Wagman RB, Ferrari S. Influence of subject discontinuation on long-term nonvertebral fracture rate in the denosumab FREEDOM Extension study. BMC Musculoskelet Disord. 2017 Apr 27;18(1):174. doi: 10.1186/s12891-017-1520-6. PMID 28449657
- [Background] Bilezikian JP, Lin CJF, Brown JP, Wang AT, Yin X, Ebeling PR, Fahrleitner-Pammer A, Franek E, Gilchrist N, Miller PD, Simon JA, Valter I, Zerbini CAF, Libanati C, Chines A. Long-term denosumab treatment restores cortical bone loss and reduces fracture risk at the forearm and humerus: analyses from the FREEDOM Extension cross-over group. Osteoporos Int. 2019 Sep;30(9):1855-1864. doi: 10.1007/s00198-019-05020-8. Epub 2019 Jun 14. PMID 31201481
- [Background] Ferrari S, Butler PW, Kendler DL, Miller PD, Roux C, Wang AT, Huang S, Wagman RB, Lewiecki EM. Further Nonvertebral Fracture Reduction Beyond 3 Years for Up to 10 Years of Denosumab Treatment. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3450-3461. doi: 10.1210/jc.2019-00271. PMID 31125092
- [Background] Ferrari S, Libanati C, Lin CJF, Brown JP, Cosman F, Czerwinski E, de Gregomicronrio LH, Malouf-Sierra J, Reginster JY, Wang A, Wagman RB, Lewiecki EM. Relationship Between Bone Mineral Density T-Score and Nonvertebral Fracture Risk Over 10 Years of Denosumab Treatment. J Bone Miner Res. 2019 Jun;34(6):1033-1040. doi: 10.1002/jbmr.3722. Epub 2019 May 29. PMID 30919997
- [Background] Broadwell A, Chines A, Ebeling PR, Franek E, Huang S, Smith S, Kendler D, Messina O, Miller PD. Denosumab Safety and Efficacy Among Participants in the FREEDOM Extension Study With Mild to Moderate Chronic Kidney Disease. J Clin Endocrinol Metab. 2021 Jan 23;106(2):397-409. doi: 10.1210/clinem/dgaa851. PMID 33211870
- [Background] Cosman F, Huang S, McDermott M, Cummings SR. Multiple Vertebral Fractures After Denosumab Discontinuation: FREEDOM and FREEDOM Extension Trials Additional Post Hoc Analyses. J Bone Miner Res. 2022 Nov;37(11):2112-2120. doi: 10.1002/jbmr.4705. Epub 2022 Oct 12. PMID 36088628
- [Derived] Bone HG, Chapurlat R, Brandi ML, Brown JP, Czerwinski E, Krieg MA, Mellstrom D, Radominski SC, Reginster JY, Resch H, Ivorra JA, Roux C, Vittinghoff E, Daizadeh NS, Wang A, Bradley MN, Franchimont N, Geller ML, Wagman RB, Cummings SR, Papapoulos S. The effect of three or six years of denosumab exposure in women with postmenopausal osteoporosis: results from the FREEDOM extension. J Clin Endocrinol Metab. 2013 Nov;98(11):4483-92. doi: 10.1210/jc.2013-1597. Epub 2013 Aug 26. PMID 23979955
- [Derived] Papapoulos S, Chapurlat R, Libanati C, Brandi ML, Brown JP, Czerwinski E, Krieg MA, Man Z, Mellstrom D, Radominski SC, Reginster JY, Resch H, Roman Ivorra JA, Roux C, Vittinghoff E, Austin M, Daizadeh N, Bradley MN, Grauer A, Cummings SR, Bone HG. Five years of denosumab exposure in women with postmenopausal osteoporosis: results from the first two years of the FREEDOM extension. J Bone Miner Res. 2012 Mar;27(3):694-701. doi: 10.1002/jbmr.1479. PMID 22113951
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an extension study open to participants who had completed core study 20030216 (NCT00089791). The study was conducted at 178 centers in North America, South America, Europe, Australia, and New Zealand. Participants were enrolled from 7 August 2007 to 20 June 2008.
Pre-assignment Details: All participants received open-label denosumab during this study. Results are reported by the Study 20030216 randomized treatment groups (placebo versus denosumab).
Groups:
- Placebo / Denosumab: Participants who were randomized to placebo in the core study received a 60 mg subcutaneous injection of denosumab every 6 months for up to seven years in the extension study.
- Denosumab / Denosumab: Participants who were randomized to denosumab in the core study received a 60 mg subcutaneous injection of denosumab every 6 months for up to seven years in the extension study (total of 10 years treatment).
Period: Overall Study
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Started | 2207 | 2343
Received Treatment | 2206 | 2343
Completed | 1283 | 1343
Not Completed | 924 | 1000
Not completed — Withdrawal by Subject | 399 | 427
Not completed — Other | 181 | 198
Not completed — Adverse Event | 122 | 155
Not completed — Death | 101 | 110
Not completed — Lost to Follow-up | 73 | 61
Not completed — Non-compliance | 20 | 13
Not completed — Physician Decision | 14 | 13
Not completed — Requirement for Alternative Therapy | 4 | 14
Not completed — Protocol Deviation | 6 | 5
Not completed — Ineligibility Determined | 3 | 4
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab | Total
Number analyzed (Participants) | 2207 | 2343 | 4550
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (5.1) | 74.9 (5.0) | 74.8 (5.0)
Age, Customized [Number; unit: participants]
  60 - 64 years | 58 | 49 | 107
  65 - 69 years | 326 | 320 | 646
  70 - 74 years | 672 | 716 | 1388
  ≥ 75 years | 1151 | 1258 | 2409
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2207 | 2343 | 4550
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 2063 | 2169 | 4232
  Black | 16 | 19 | 35
  Hispanic or Latino | 121 | 145 | 266
  Asian | 2 | 3 | 5
  Japanese | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 1 | 2 | 3
Bone Mineral Density T-score [Mean (Standard Deviation); unit: T-score] — The T-score is the bone mineral density (BMD) at the site when compared to that of a healthy thirty-year-old.
  Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman.
  T-score
    Lumbar spine | -2.81 (0.75) | -2.14 (0.80) | -2.47 (0.84)
    Total hip | -1.93 (0.80) | -1.50 (0.79) | -1.71 (0.83)
    Femoral neck | -2.17 (0.72) | -1.83 (0.75) | -1.99 (0.75)
Bone Mineral Density T-score at Study 20030216 Baseline [Mean (Standard Deviation); unit: T-score]
  Lumbar spine | -2.84 (0.68) | -2.83 (0.67) | -2.83 (0.68)
  Total hip | -1.85 (0.79) | -1.85 (0.79) | -1.85 (0.79)
  Femoral neck | -2.11 (0.71) | -2.11 (0.71) | -2.11 (0.71)
Any Historical Fracture at Age ≥ 55 Years [Number; unit: participants] | 1089 | 1133 | 2222

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: A serious adverse event (SAE) is defined as an adverse event that: • is fatal • is life threatening • requires in-patient hospitalization or prolongation of existing hospitalization • results in persistent or significant disability/incapacity • is a congenital anomaly/birth defect • is other significant medical hazard. Treatment-related adverse events includes only events for which the investigator indicated there was a reasonable possibility they may have been caused by study drug. The following were classified as adverse events of interest (events that are considered to be identified or potential risks of denosumab treatment): positively adjudicated osteonecrosis of the jaw, positively adjudicated atypical femoral fracture, hypocalcemia, adverse events potentially related to hypersensitivity, serious infection (including bacterial cellulitis), malignancy, cardiac disorders, vascular disorders, fracture healing complications, eczema, acute pancreatitis, and musculoskeletal pain.
Time Frame: 84 months
Population: All participants who received at least one dose of denosumab.
Measure: Number; unit: participants
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 2206 | 2343
participants
  Any adverse event (AE) | 2070 | 2173
  Serious adverse event | 945 | 1014
  Fatal adverse event | 101 | 108
  AE leading to study discontinuation | 145 | 173
  AE leading to discontinuation of denosumab | 184 | 216
  Treatment-related adverse events (TRAE) | 185 | 188
  Serious treatment-related adverse events | 26 | 28
  Fatal treatment-related adverse events | 1 | 0
  TRAE leading to study discontinuation | 16 | 9
  TRAE leading to discontinuation of denosumab | 30 | 25
  Positively adjudicated osteonecrosis of the jaw | 6 | 7
  Positively adjudicated atypical femoral fracture | 1 | 1
  Hypocalcaemia | 10 | 6
  AEs potentially related to hypersensitivity | 260 | 280
  Serious infections | 161 | 185
  Serious bacterial cellulitis | 7 | 12
  Malignancy | 227 | 237
  Cardiac disorders | 449 | 492
  Vascular disorders | 693 | 732
  Fracture healing complications | 0 | 1
  Eczema | 99 | 115
  Acute pancreatitis | 4 | 8
  Musculoskeletal pain | 1125 | 1206

2. Primary Outcome: Number of Participants With Laboratory Toxicities of Grade ≥ 3
Description: Laboratory toxicity grading was based on Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Grade 3 indicates severe toxicity and Grade 4 indicates life-threatening toxicity.
Time Frame: 84 months
Population: All participants who received at least 1 dose of denosumab
Measure: Number; unit: participants
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 2206 | 2343
participants
  Low sodium - Grade 3 | 28 | 25
  Low sodium - Grade 4 | 1 | 0
  High potassium - Grade 3 | 9 | 11
  High potassium - Grade 4 | 0 | 3
  Low potassium - Grade 3 | 7 | 7
  Low magnesium - Grade 3 | 1 | 1
  Low magnesium - Grade 4 | 0 | 1
  High calcium - Grade 3 | 2 | 3
  High calcium - Grade 4 | 0 | 2
  High corrected calcium - Grade 3 | 2 | 3
  High corrected calcium - Grade 4 | 0 | 2
  Low phosphorus - Grade 3 | 3 | 1
  High Creatinine - Grade 3 | 0 | 1
  High aspartate amino transferase (AST) - Grade 3 | 5 | 11
  High aspartate amino transferase (AST) - Grade 4 | 1 | 0
  High alanine amino transferase (ALT) - Grade 3 | 8 | 10
  High alanine amino transferase (ALT) - Grade 4 | 1 | 0
  High total bilirubin - Grade 3 | 2 | 3
  Low albumin - Grade 3 | 0 | 1
  High glucose - Grade 3 | 35 | 37
  High glucose - Grade 4 | 0 | 1
  Low glucose - Grade 3 | 4 | 1
  Low glucose - Grade 4 | 1 | 1
  Low hemoglobin - Grade 3 | 6 | 4
  Low platelets - Grade 3 | 3 | 7
  Low platelets - Grade 4 | 2 | 4
  Low white blood cells - Grade 3 | 5 | 7
  Low white blood cells - Grade 4 | 0 | 1
  Low lymphocytes - Grade 3 | 17 | 16
  Low lymphocytes - Grade 4 | 2 | 1

3. Primary Outcome: Number of Participants With Antibodies to Denosumab
Time Frame: Every 12 months through Month 84
Population: All participants who received at least 1 dose of denosumab
Measure: Number; unit: participants
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 2206 | 2343
participants | 1 | 0

4. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density by Visit
Description: Lumbar spine bone mineral density (BMD) was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline (of extension study) and months 12, 24, 36, 60 and 84
Population: Participants with an Extension Study baseline and at least 1 post-baseline DXA BMD measurement. "n" indicates the number of participants with available data at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 2089 | 2210
percent change
  Month 12 (n = 2040, 2168) | 5.2 [5.0 to 5.3] | 2.0 [1.8 to 2.2]
  Month 24 (n = 1935, 2061) | 7.7 [7.5 to 7.9] | 3.5 [3.4 to 3.7]
  Month 36 (n = 1497, 1607) | 9.4 [9.1 to 9.6] | 4.9 [4.7 to 5.1]
  Month 60 (n = 1472, 1567) | 13.0 [12.7 to 13.3] | 7.9 [7.6 to 8.2]
  Month 84 (n = 1223, 1264) | 16.5 [16.1 to 16.9] | 10.8 [10.4 to 11.2]

5. Secondary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density by Visit
Description: Total hip bone mineral density was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline (of extension study) and months 12, 24, 36, 60 and 84
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 2089 | 2210
percent change
  Month 12 (n = 2029, 2160) | 3.0 [2.8 to 3.1] | 0.8 [0.7 to 0.9]
  Month 24 (n = 1918, 2045) | 4.1 [4.0 to 4.2] | 1.4 [1.3 to 1.5]
  Month 36 (n = 1475, 1591) | 4.9 [4.7 to 5.0] | 1.8 [1.7 to 2.0]
  Month 60 (n = 1439, 1538) | 6.2 [6.0 to 6.4] | 2.6 [2.4 to 2.8]
  Month 84 (n = 1200, 1232) | 7.4 [7.1 to 7.6] | 3.4 [3.2 to 3.7]

6. Secondary Outcome: Percent Change From Baseline in Femoral Neck Bone Mineral Density by Visit
Description: Femoral neck bone mineral density was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline (of extension study) and months 12, 24, 36, 60 and 84
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 2089 | 2210
percent change
  Month 12 (n = 2029, 2160) | 2.1 [1.9 to 2.3] | 0.8 [0.7 to 1.0]
  Month 24 (n = 1918, 2045) | 3.2 [3.1 to 3.4] | 1.2 [1.0 to 1.4]
  Month 36 (n = 1475, 1591) | 4.0 [3.8 to 4.3] | 1.7 [1.5 to 1.9]
  Month 60 (n = 1439, 1538) | 5.7 [5.4 to 5.9] | 2.8 [2.6 to 3.1]
  Month 84 (n = 1200, 1232) | 7.1 [6.8 to 7.4] | 3.8 [3.5 to 4.2]

7. Secondary Outcome: Percent Change From Baseline in 1/3 Radius Bone Mineral Density by Visit
Description: 1/3 radius bone mineral density was measured in a subset of participants by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center.
Time Frame: Baseline (of extension study) and months 12, 24, 36, 60 and 84
Population: Participants in the DXA substudy with an Extension Study baseline and at least 1 post-baseline DXA BMD measurement. "n" indicates the number of participants with available data at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 449 | 467
percent change
  Month 12 (n = 114, 134) | 0.3 [-0.2 to 0.9] | 0.6 [0.1 to 1.2]
  Month 24 (n = 108, 127) | 0.2 [-0.4 to 0.9] | 0.2 [-0.4 to 0.8]
  Month 36 (n = 73, 93) | 1.3 [0.5 to 2.0] | 0.6 [-0.1 to 1.3]
  Month 60 (n = 59, 84) | 1.8 [0.9 to 2.7] | 1.4 [0.6 to 2.2]
  Month 84 (n = 39, 56) | 2.2 [0.9 to 3.6] | 1.0 [-0.1 to 2.2]

8. Secondary Outcome: Percent Change From Study 20030216 Baseline in Lumbar Spine Bone Mineral Density by Visit
Description: Lumbar spine bone mineral density was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center. Measurements at some time points during the core study 20030216 were only taken in a subset of participants.
Time Frame: Study 20030216 baseline and extension study months 12, 24, 36, 60 and 84
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 2089 | 2210
percent change
  Month 12 (n = 2030, 2148) | 5.9 [5.6 to 6.1] | 11.9 [11.7 to 12.2]
  Month 24 (n = 1924, 2041) | 8.4 [8.1 to 8.7] | 13.7 [13.4 to 13.9]
  Month 36 (n = 1487, 1589) | 10.1 [9.8 to 10.4] | 15.2 [14.9 to 15.5]
  Month 60 (n = 1464, 1551) | 13.8 [13.4 to 14.1] | 18.4 [18.1 to 18.8]
  Month 84 (n = 1216, 1251) | 17.3 [16.8 to 17.8] | 21.7 [21.2 to 22.2]

9. Secondary Outcome: Percent Change From Study 20030216 Baseline in Total Hip BMD by Visit
Description: Total hip bone mineral density was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center. Measurements at some time points during the core study 20030216 were only taken in a subset of participants.
Time Frame: Study 20030216 baseline and extension study months 12, 24, 36, 60 and 84
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 2089 | 2210
percent change
  Month 12 (n = 2006, 2132) | 1.7 [1.6 to 1.9] | 6.4 [6.3 to 6.6]
  Month 24 (n = 1895, 2017) | 2.9 [2.7 to 3.0] | 7.1 [6.9 to 7.2]
  Month 36 (n = 1457, 1567) | 3.6 [3.4 to 3.8] | 7.5 [7.3 to 7.7]
  Month 60 (n = 1424, 1518) | 4.9 [4.7 to 5.2] | 8.4 [8.1 to 8.6]
  Month 84 (n = 1189, 1215) | 6.1 [5.8 to 6.4] | 9.2 [8.9 to 9.5]

10. Secondary Outcome: Percent Change From Study 20030216 Baseline in Femoral Neck BMD by Visit
Description: Femoral neck bone mineral density was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center. Measurements at some time points during the core study 20030216 were only taken in a subset of participants.
Time Frame: Study 20030216 baseline and extension study months 12, 24, 36, 60 and 84
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 2089 | 2210
percent change
  Month 12 (n = 2006, 2132) | 1.4 [1.2 to 1.7] | 5.8 [5.6 to 6.0]
  Month 24 (n = 1895, 2017) | 2.6 [2.3 to 2.8] | 6.2 [6.0 to 6.5]
  Month 36 (n = 1457, 1567) | 3.4 [3.1 to 3.6] | 6.7 [6.5 to 7.0]
  Month 60 (n = 1424, 1518) | 5.0 [4.7 to 5.3] | 7.9 [7.6 to 8.2]
  Month 84 (n = 1189, 1215) | 6.4 [6.0 to 6.8] | 9.0 [8.6 to 9.4]

11. Secondary Outcome: Percent Change From Study 20030216 Baseline in 1/3 Radius BMD by Visit
Description: 1/3 radius BMD was measured by dual x-ray absorptiometry (DXA). DXA scans were analyzed by a central imaging center. Measurements at some time points during the core study 20030216 were only taken in a subset of participants.
Time Frame: Study 20030216 baseline and extension study months 12, 24, 36, 60, and 84
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 449 | 467
percent change
  Month 12 (n = 113, 133) | -1.0 [-1.7 to -0.3] | 2.6 [1.9 to 3.2]
  Month 24 (n = 107, 127) | -1.2 [-1.9 to -0.4] | 2.1 [1.4 to 2.8]
  Month 36 (n = 73, 92) | -0.2 [-1.1 to 0.7] | 2.4 [1.6 to 3.2]
  Month 60 (n = 59, 83) | 0.3 [-0.7 to 1.3] | 3.3 [2.4 to 4.2]
  Month 84 (n = 39, 56) | 0.6 [-0.8 to 2.1] | 2.8 [1.6 to 4.1]

12. Secondary Outcome: Number of Participants With New Vertebral Fractures
Description: A new vertebral fracture, assessed by lateral spine X-ray using Genant semiquantitative scoring method, was identified as an ≥ 1 grade increase from the previous grade of 0 in any vertebra from T4 to L4, excluding any fracture associated with high trauma severity or a pathologic fracture.
Time Frame: 84 months
Population: All participants enrolled in the extension study who have vertebral X-ray assessment at the extension baseline and at least 1 post-extension baseline visit.
Measure: Number; unit: participants
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 1991 | 2116
participants | 145 | 149

13. Secondary Outcome: Number of Participants With Non-Vertebral Fractures
Description: Non-vertebral fractures (osteoporotic) were defined as a fracture present on a copy of radiographs or other diagnostic images such as computerized tomography (CT) or magnetic resonance imaging (MRI) confirming the fracture, and/or documented in a copy of the radiology report, surgical report, or discharge summary, excluding skull, facial, mandible, cervical vertebrae, thoracic vertebrae, lumbar vertebrae, metacarpus, finger phalanges, and toe phalanges. In addition, fractures associated with high trauma severity or pathologic fractures were excluded.
Time Frame: 84 months
Population: All enrolled participants
Measure: Number; unit: participants
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 2207 | 2343
participants | 219 | 172

14. Secondary Outcome: Percent Change From Baseline in C-Telopeptide 1 (CTX-1) by Visit
Description: Bone turnover markers were collected in a subset of participants who participated in the 20030216 Bone Marker sub-study and in new participants continuing beyond month 24 who were not previously in the Bone Turnover Markers sub-study.
Time Frame: Baseline (of extension study), day 10, and months 6, 12, 24, 36, 48, 60, 72, and 84
Population: Participants who received at least 1 dose of denosumab and enrolled in the bone turnover marker substudy at screening or Month 24 in Study 20060289. "n" indicates the number of participants with available data at each time point.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 318 | 342
percent change
  Day 10 (n = 26, 47) | -90 [-93 to -85] | -72 [-86 to -47]
  Month 6 (n = 30, 56) | -85 [-91 to -73] | -26 [-63 to 1]
  Month 12 (n = 27, 56) | -75 [-90 to -54] | -13 [-37 to 24]
  Month 24 (n = 27, 47) | -67 [-84 to -29] | 10 [-27 to 55]
  Month 36 (n = 68, 81) | -59 [-84 to -28] | 2 [-32 to 68]
  Month 48 (n = 62, 75) | -58 [-84 to -12] | 0 [-46 to 56]
  Month 60 (n = 59, 70) | -65 [-90 to -19] | 0 [-47 to 83]
  Month 72 (n = 56, 62) | -60 [-85 to -16] | -1 [-47 to 76]
  Month 84 (n = 41, 41) | -64 [-86 to -28] | -6 [-26 to 68]

15. Secondary Outcome: Percent Change From Baseline in Procollagen Type 1 N-telopeptide (P1NP) by Visit
Description: Bone turnover markers were collected in a subset of participants who participated in the 20030216 Bone Marker sub-study and in new sparticipants continuing beyond month 24 who were not previously in the Bone Turnover Markers sub-study.
Time Frame: Baseline (of extension study), day 10, and months 6, 12, 24, 36, 48, 60, 72, and 84
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 318 | 342
percent change
  Day 10 (n = 30, 51) | 6 [-5 to 30] | 14 [-1 to 25]
  Month 6 (n = 30, 53) | -71 [-78 to -62] | -23 [-50 to -2]
  Month 12 (n = 26, 56) | -67 [-76 to -57] | 7 [-15 to 30]
  Month 24 (n = 27, 47) | -63 [-77 to -41] | 11 [-17 to 42]
  Month 36 (n = 69, 83) | -57 [-67 to -29] | 29 [-6 to 91]
  Month 48 (n = 61, 73) | -60 [-70 to -41] | 8 [-21 to 49]
  Month 60 (n = 61, 71) | -54 [-72 to -35] | 30 [-6 to 67]
  Month 72 (n = 55, 64) | -50 [-60 to -36] | 44 [3 to 103]
  Month 84 (n = 48, 50) | -59 [-73 to -40] | 32 [-4 to 75]

16. Secondary Outcome: Percent Change From Study 20030216 Baseline in CTX-1 by Visit
Description: as for outcome 14
Time Frame: Study 20030216 Baseline and extension study day 10, and months 6, 12, 24, 36, 48, 60, 72, and 84
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 318 | 342
percent change
  Day 10 (n = 26, 56) | -90 [-91 to -78] | -91 [-93 to -86]
  Month 6 (n = 32, 72) | -83 [-90 to -72] | -77 [-87 to -49]
  Month 12 (n = 27, 65) | -77 [-91 to -45] | -63 [-87 to -11]
  Month 24 (n = 28, 60) | -65 [-80 to -24] | -53 [-82 to 0]
  Month 36 (n = 289, 313) | -71 [-88 to -40] | -52 [-86 to -4]
  Month 48 (n = 274, 290) | -70 [-88 to -36] | -61 [-85 to -24]
  Month 60 (n = 268, 276) | -67 [-88 to -25] | -53 [-86 to -18]
  Month 72 (n = 243, 248) | -69 [-88 to -32] | -59 [-86 to -21]
  Month 84 (n = 217, 216) | -63 [-88 to -19] | -53 [-84 to -12]

17. Secondary Outcome: Percent Change From Study 20030216 Baseline in P1NP by Visit
Description: as for outcome 14
Time Frame: Study 20030216 Baseline and extension study day 10, and months 6, 12, 24, 36, 48, 60, 72, and 84
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 318 | 342
percent change
  Day 10 (n = 30, 51) | 9 [-14 to 34] | -59 [-74 to -22]
  Month 6 (n = 32, 57) | -74 [-80 to -67] | -75 [-80 to -55]
  Month 12 (n = 26, 56) | -74 [-79 to -51] | -63 [-76 to -36]
  Month 24 (n = 28, 51) | -67 [-75 to -51] | -56 [-72 to -30]
  Month 36 (n = 70, 83) | -59 [-75 to -37] | -60 [-71 to -40]
  Month 48 (n = 61, 73) | -67 [-75 to -46] | -63 [-77 to -42]
  Month 60 (n = 61, 71) | -62 [-75 to -42] | -55 [-74 to -30]
  Month 72 (n = 56, 67) | -62 [-71 to -35] | -55 [-70 to -27]
  Month 84 (n =49, 53) | -68 [-78 to -56] | -57 [-74 to -38]

18. Secondary Outcome: Percent Change From Baseline in Albumin-adjusted Serum Calcium at Day 10
Time Frame: Baseline (of extension study) and day 10
Population: Participants who had a calcium corrected by albumin measurement within the Day 10 visit window up to May 31, 2008.
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 2027 | 2154
percent change | -3.1 [-6.1 to 0.0] | -2.0 [-5.1 to 1.1]

19. Secondary Outcome: Serum Denosumab Concentration
Description: Serum concentrations of denosumab were measured by a validated conventional sandwich enzyme-linked immunosorbent assay (ELISA). The lower limit of quantification (LLOQ) was 0.8 ng/mL. Values of 0 in the table below indicate data below the lower limit of quantification.
Time Frame: Baseline (pre-dose in extension study), day 10, and Months 3, 4 and 6 (pre-dose)
Population: Participants who participated in the Study 20030216 PK substudy, for whom dosing information was not missing and for whom sampling was within 14 days of specified sampling times.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 97 | 113
ng/mL
  Baseline (n = 97, 113) | 0 (0) | 113 (107)
  Day 10 (n = 92, 106) | 5890 (2010) | 6010 (2530)
  Month 3 (n = 81, 92) | 1000 (560) | 1190 (690)
  Month 4 (n = 87, 104) | 429 (378) | 554 (480)
  Month 6 (n = 87, 103) | 20.8 (61.7) | 66.0 (147.2)

20. Secondary Outcome: Bone Histomorphometry: Cancellous Bone Volume
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. Cancellous (trabecular) bone volume is the percent of the total marrow cavity that is occupied by cancellous bone (both mineralized and non-mineralized) measured by quantitative histomorphometry.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available cancellous bone volume data.
Measure: Mean (Standard Deviation); unit: percentage of total bone tissue volume
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
percentage of total bone tissue volume
  Month 24 (n = 13, 25) | 15.253 (6.065) | 14.640 (6.979)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 16.358 (4.438)

21. Secondary Outcome: Bone Histomorphometry: Trabecular Number
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. Trabecular number is the number of trabeculae present per lineal mm and is calculated as trabecular bone volume/trabecular thickness. Trabecular number is a measure of trabecular connectivity and decreases with bone loss.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available trabecular number data.
Measure: Mean (Standard Deviation); unit: 1/mm
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
1/mm
  Month 24 (n = 13, 25) | 1.005 (0.242) | 0.904 (0.243)
  Month 24 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 1.235 (0.254)

22. Secondary Outcome: Bone Histomorphometry: Trabecular Separation
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. Trabecular separation is the mean distance between trabeculae (measured by integrated computer graphics). Trabecular separation increases with trabecular bone loss.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available trabecular separation data.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
μm
  Month 24 (n = 13, 25) | 919.693 (358.238) | 1033.416 (352.259)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 708.669 (171.782)

23. Secondary Outcome: Bone Histomorphometry: Trabecular Thickness
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. Mean trabecular thickness is a measure of trabecular structure and is calculated as the reciprocal of total bone (trabecular) surfaces. Trabecular thickness is reduced by aging and osteoporosis.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available trabecular thickness data.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
μm
  Month 24 (n = 13, 25) | 153.878 (51.859) | 156.335 (48.567)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 132.965 (28.064)

24. Secondary Outcome: Bone Histomorphometry: Cortical Width
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. Cortical width is the average width of both inner and outer cortices.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available cortical width data.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 45
μm
  Month 24 (n = 13, 28) | 622.22 (246.70) | 707.69 (237.97)
  Month 84 (n = 0, 21) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 786.19 (279.81)

25. Secondary Outcome: Bone Histomorphometry: Cancellous Bone Volume by TRAP Histomorphometry
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. Cancellous (trabecular) bone volume is the percent of the total marrow cavity that is occupied by cancellous bone (both mineralized and non-mineralized) measured by tartrate-resistant acid phosphatase (TRAP) staining histomorphometry.
Time Frame: Month 24 and month 84
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: percentage of total bone tissue volume
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
percentage of total bone tissue volume
  Month 24 (n = 13, 25) | 16.678 (7.270) | 15.606 (6.986)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 17.631 (4.387)

26. Secondary Outcome: Bone Histomorphometry: Surface Density
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. Surface density is calculated by total bone (trabecular) surfaces / total tissue volume.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available surface density data.
Measure: Mean (Standard Deviation); unit: mm²/mm³
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
mm²/mm³
  Month 24 (n = 13, 25) | 2.009 (0.486) | 1.807 (0.486)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 2.472 (0.506)

27. Secondary Outcome: Bone Histomorphometry: Osteoblast - Osteoid Interface
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. Osteoblast - osteoid interface is calculated as osteoblast surface / osteoid surface * 100.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available osteoblast - osteoid interface data.
Measure: Mean (Standard Deviation); unit: percentage of osteoid surface
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
percentage of osteoid surface
  Month 24 (n = 13, 25) | 22.124 (34.879) | 17.813 (28.381)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 5.951 (15.223)

28. Secondary Outcome: Bone Histomorphometry: Osteoid Surface
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. Osteoid surface is the percent of bone surface covered in osteoid.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available osteoid surface data.
Measure: Mean (Standard Deviation); unit: percentage of total bone surface
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
percentage of total bone surface
  Month 24 (n = 13, 25) | 0.915 (1.382) | 0.982 (2.489)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.421 (1.068)

29. Secondary Outcome: Bone Histomorphometry: Osteoid Thickness
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. Osteoid thickness (width) is the mean thickness of osteoid seams on cancellous surfaces. Osteoid thickness is normally <12.5 µm. Increased osteoid thickness suggests abnormal mineralization (osteomalacia).
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available osteoid thickness data.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
μm
  Month 24 (n = 13, 25) | 5.139 (3.261) | 4.548 (4.973)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 4.108 (3.476)

30. Secondary Outcome: Bone Histomorphometry: Wall Thickness
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. Wall thickness is the average thickness of trabecular bone structural units (BSU) and is used to assess the overall balance between resorption and formation.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available wall thickness data.
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
μm
  Month 24 (n = 13, 25) | 43.11 (6.08) | 49.74 (10.51)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 39.59 (7.49)

31. Secondary Outcome: Bone Histomorphometry: Eroded Surface/Bone Surface
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  Eroded surface/bone surface is the percentage of bone surface occupied by eroded (resorption) cavities (Howships lacunae), with or without osteoclasts.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available eroded surface/bone surface data.
Measure: Mean (Standard Deviation); unit: percentage of bone surface
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
percentage of bone surface
  Month 24 (n = 13, 25) | 0.414 (0.701) | 0.328 (0.613)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.511 (0.579)

32. Secondary Outcome: Bone Histomorphometry: Osteoclast Number - Length Based
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  Osteoclast number was measured by quantitative histomorphometry and is expressed per mm of bone.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available osteoclast number data.
Measure: Mean (Standard Deviation); unit: 1/mm
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
1/mm
  Month 24 (n = 13, 25) | 0.086 (0.119) | 0.107 (0.198)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.074 (0.101)

33. Secondary Outcome: Bone Histomorphometry: Osteoclast Number - Surface Based
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  Osteoclast number was measured by quantitative histomorphometry and is expressed per 100 mm of bone surface area.
Time Frame: Month 24 and month 84
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 1/100 mm
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
1/100 mm
  Month 24 (n = 13, 25) | 8.6 (11.9) | 10.7 (19.8)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 7.4 (10.1)

34. Secondary Outcome: Bone Histomorphometry: Osteoclast Number by TRAP - Length Based
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  Osteoclast number was measured using TRAP staining and is expressed per mm of bone.
Time Frame: Month 24 and month 84
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 1/mm
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
1/mm
  Month 24 (n = 13, 25) | 0.096 (0.134) | 0.110 (0.185)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.077 (0.107)

35. Secondary Outcome: Bone Histomorphometry: Osteoclast Number by TRAP - Surface Based
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  Osteoclast number was measured using TRAP staining and is expressed per 100 mm of bone surface.
  Da
Time Frame: Month 24 and month 84
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: 1/100 mm
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
1/100 mm
  Month 24 (n = 13, 25) | 9.6 (13.4) | 11.0 (18.5)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 7.7 (10.7)

36. Secondary Outcome: Bone Histomorphometry: Single-label Surface
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  A double tetracycline labeling procedure was used to allow visualization and quantification of sites of new bone formation. Tetracycline was given for two periods of 3 days separated by 14 days where no tetracycline was taken. A single label is deposited if formation either started or ended during the interval between the uses of the two courses of tetracycline administration. Single-label surface is expressed as a percentage of total bone surface.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available single-label surface data.
Measure: Mean (Standard Deviation); unit: percentage of bone surface
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 5 | 20
percentage of bone surface
  Month 24 (n = 5, 10) | 0.304 (0.302) | 0.643 (0.661)
  Month 84 (n = 0, 10) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.611 (0.726)

37. Secondary Outcome: Bone Histomorphometry: Double-label Surface
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  A double tetracycline labeling procedure was used to allow visualization and quantification of sites of new bone formation. Tetracycline was given for two periods of 3 days separated by 14 days where no tetracycline was taken. The presence of double labels indicates that normal bone mineralization was actively occurring over the entire labeling interval. Double-label surface is expressed as a percentage of total bone surface.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available double-label surface data.
Measure: Mean (Standard Deviation); unit: percentage of bone surface
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 5 | 20
percentage of bone surface
  Month 24 (n = 5, 10) | 0.258 (0.207) | 0.356 (0.295)
  Month 84 (n = 0, 10) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.106 (0.237)

38. Secondary Outcome: Bone Histomorphometry: Mineralizing Surface
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  A double tetracycline labeling procedure was used to allow visualization and quantification of sites of new bone formation. Tetracycline was given for two periods of 3 days separated by 14 days where no tetracycline was taken. Total mineralizing surfaces (MS) include all double and half of single-labeled surfaces. MS is expressed as a percentage of total bone surface.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available mineralizing surface data.
Measure: Mean (Standard Deviation); unit: percentage of bone surface
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 5 | 20
percentage of bone surface
  Month 24 (n = 5, 10) | 0.406 (0.323) | 0.681 (0.453)
  Month 84 (n = 0, 10) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.412 (0.458)

39. Secondary Outcome: Bone Histomorphometry: Mineral Apposition Rate
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  A double tetracycline labeling procedure was used to allow visualization and quantification of sites of new bone formation. Tetracycline was given for two periods of 3 days separated by 14 days where no tetracycline was taken. The mineral apposition rate (MAR) is the avarage rate at which new bone mineral is being added on any actively forming surface. MAR is calculated as the average distance between visible labels, divided by the labeling interval.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available mineral apposition rate data.
Measure: Mean (Standard Deviation); unit: μm/day
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 5 | 20
μm/day
  Month 24 (n = 5, 10) | 0.616 (0.219) | 0.722 (0.573)
  Month 84 (n = 0, 10) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.394 (0.233)

40. Secondary Outcome: Bone Histomorphometry: Adjusted Apposition Rate
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  A double tetracycline labeling procedure was used to allow visualization and quantification of sites of new bone formation. Tetracycline was given for two periods of 3 days separated by 14 days where no tetracycline was taken. The mineral apposition rate (MAR) is the average rate at which new bone mineral is being added on any actively forming surface. Adjusted MAR is calculated as: (average distance between visible labels / labeling interval) * (total mineralizing surface/total bone surface).
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available adjusted apposition rate data.
Measure: Mean (Standard Deviation); unit: μm/day
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 5 | 19
μm/day
  Month 24 (n = 5, 9) | 0.394 (0.471) | 0.517 (0.537)
  Month 84 (n = 0, 10) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.818 (1.207)

41. Secondary Outcome: Bone Histomorphometry: Bone Formation Rate - Surface Based
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  A double tetracycline labeling procedure was used to allow visualization and quantification of sites of new bone formation. Tetracycline was given for two periods of 3 days separated by 14 days where no tetracycline was taken. Bone formation rate - surface based is the calculated rate at which cancellous bone surface is being replaced annually, derived from the Mineral Appositional Rate * 365 * (relative mineralizing surface / total bone surface).
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available bone formation rate data.
Measure: Mean (Standard Deviation); unit: μm³/μm²/year
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 5 | 20
μm³/μm²/year
  Month 24 (n = 5, 10) | 0.898 (0.706) | 2.153 (2.468)
  Month 84 (n = 0, 10) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.691 (0.868)

42. Secondary Outcome: Bone Histomorphometry: Bone Formation Rate - Volume Based
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  A double tetracycline labeling procedure was used to allow visualization and quantification of sites of new bone formation. Tetracycline was given for two periods of 3 days separated by 14 days where no tetracycline was taken. Bone formation rate - volume based is the calculated rate at which cancellous bone volume is being replaced annually, derived from the Mineral Appositional Rate * 365 * (relative mineralizing surface / total bone volume).
Time Frame: Month 24 and month 84
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: percent of bone volume per year
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 5 | 20
percent of bone volume per year
  Month 24 (n = 5, 10) | 1.454 (1.265) | 3.162 (3.773)
  Month 84 (n = 0, 10) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 1.071 (1.308)

43. Secondary Outcome: Bone Histomorphometry: Formation Period
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  A double tetracycline labeling procedure was used to allow visualization and quantification of sites of new bone formation. Tetracycline was given for two periods of 3 days separated by 14 days where no tetracycline was taken. Formation period (FP) is the mean time required to rebuild a new bone structural unit or osteon from the cement line back to the bone surface at a single location, and is given by wall width / adjusted apposition rate.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available formation period data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 5 | 20
days
  Month 24 (n = 5, 10) | 593.5 (996.8) | 287.3 (391.5)
  Month 84 (n = 0, 10) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 229.7 (512.0)

44. Secondary Outcome: Bone Histomorphometry: Activation Frequency
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  A double tetracycline labeling procedure was used to allow visualization and quantification of sites of new bone formation. Tetracycline was given for two periods of 3 days separated by 14 days where no tetracycline was taken. The average time that it takes for a new remodeling cycle to begin on any point on a cancellous surface is called the activation frequency. Activation frequency is calculated as the bone formation rate / wall width.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available activation frequency data.
Measure: Mean (Standard Deviation); unit: /year
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 5 | 20
/year
  Month 24 (n = 5, 10) | 0.022 (0.019) | 0.045 (0.049)
  Month 84 (n = 0, 10) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.014 (0.024)

45. Secondary Outcome: Bone Histomorphometry: Osteoid Volume
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry.
  Osteoid volume is the percentage of a given volume of bone tissue that consists of unmineralized bone (osteoid).
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available osteoid volume data.
Measure: Mean (Standard Deviation); unit: percentage of total bone tissue
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 41
percentage of total bone tissue
  Month 24 (n = 13, 25) | 0.108 (0.193) | 0.146 (0.382)
  Month 84 (n = 0, 19) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 0.048 (0.133)

46. Secondary Outcome: Bone Histomorphometry: Mineralization Lag Time
Description: Bone biopsy samples were prepared according to standard procedures for bone histomorphometry. A double tetracycline labeling procedure was used to allow visualization and quantification of sites of new bone formation. Tetracycline was given for two periods of 3 days separated by 14 days where no tetracycline was taken.
  Mineralization lag time is the average time interval between osteoid formation and its subsequent mineralization and is calculated by dividing the osteoid width by the apposition rate.
Time Frame: Month 24 and month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, had at least 1 bone biopsy evaluable for histomorphometry at extension month 24 or extension month 84 and with available mineralization lag time data.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 5 | 20
days
  Month 24 (n = 5, 10) | 84.9 (136.8) | 54.3 (76.1)
  Month 84 (n = 0, 10) | NA (NA) — No participants in this arm had a bone biopsy evaluable for histomorphometry at month 84 | 52.3 (114.5)

47. Secondary Outcome: Bone Histology at Month 24
Description: Bone biopsy samples were prepared according to standard procedures for bone histology to determine if there were any histological abnormalities in the bone. Results are reported for the number of biopsies with normal bone micro-architecture: normal lamellar bone, normal mineralization, and osteoid, and biopsies with abnormal bone histology: osteomalacia, marrow fibrosis, or woven bone.
Time Frame: Month 24
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, and had at least 1 bone biopsy evaluable for histology at extension month 24.
Measure: Number; unit: biopsies
Units Other Than Participants: biopsies
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 13 | 28
Number analyzed (biopsies) | 13 | 28
biopsies
  Normal lamellar bone | 13 | 28
  Normal mineralization | 13 | 28
  Osteoid | 13 | 23
  Osteomalacia | 0 | 0
  Marrow fibrosis | 0 | 0
  Woven bone | 0 | 0

48. Secondary Outcome: Bone Histology at Month 84
Description: as for outcome 47
Time Frame: Month 84
Population: Participants who enrolled in the bone biopsy substudy, received at least 1 dose of denosumab during the extension study, and had at least 1 bone biopsy evaluable for histology at extension month 84.
Measure: Number; unit: biopsies
Units Other Than Participants: biopsies
Arm/Group | Placebo / Denosumab | Denosumab / Denosumab
Number analyzed (Participants) | 0 | 22
Number analyzed (biopsies) | 0 | 22
biopsies
  Normal lamellar bone |  | 22
  Normal mineralization |  | 22
  Osteoid |  | 18
  Osteomalacia |  | 0
  Marrow fibrosis |  | 0
  Woven bone |  | 0

ADVERSE EVENTS:
Time Frame: 84 months
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Placebo/ Denosumab 60 mg Q6M: Participants who were randomized to placebo in the core study received a 60 mg subcutaneous injection of denosumab every 6 months for up to seven years.
- Denosumab/ Denosumab 60 mg Q6M: Participants who were randomized to denosumab in the core study received a 60 mg subcutaneous injection of denosumab every 6 months for up to seven years (total of 10 years treatment).
Arm/Group | Placebo/ Denosumab 60 mg Q6M | Denosumab/ Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 945/2206 | 1014/2343
Other Adverse Events (participants affected / at risk) | 1809/2206 | 1920/2343
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/ Denosumab 60 mg Q6M (N=2206) | Denosumab/ Denosumab 60 mg Q6M (N=2343)
Anaemia (Blood and lymphatic system disorders) | 11 | 11
Bone marrow oedema (Blood and lymphatic system disorders) | 2 | 1
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 8 | 18
Adams-Stokes syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 17 | 19
Angina unstable (Cardiac disorders) | 7 | 12
Aortic valve disease (Cardiac disorders) | 0 | 3
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Aortic valve stenosis (Cardiac disorders) | 4 | 3
Arrhythmia (Cardiac disorders) | 3 | 4
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 50 | 40
Atrial flutter (Cardiac disorders) | 0 | 4
Atrioventricular block (Cardiac disorders) | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 5 | 4
Atrioventricular block second degree (Cardiac disorders) | 2 | 2
Bradycardia (Cardiac disorders) | 5 | 3
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 4 | 4
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 15 | 21
Cardiac failure acute (Cardiac disorders) | 1 | 3
Cardiac failure chronic (Cardiac disorders) | 1 | 3
Cardiac failure congestive (Cardiac disorders) | 10 | 9
Cardiac fibrillation (Cardiac disorders) | 1 | 0
Cardiac valve disease (Cardiac disorders) | 0 | 2
Cardiac valve sclerosis (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2
Cardiogenic shock (Cardiac disorders) | 0 | 2
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 4 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Chronic right ventricular failure (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 9 | 17
Coronary artery insufficiency (Cardiac disorders) | 3 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 6
Extrasystoles (Cardiac disorders) | 0 | 1
Heart valve calcification (Cardiac disorders) | 2 | 0
Heart valve incompetence (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 2 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 1
Left atrial dilatation (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 2 | 3
Mitral valve disease (Cardiac disorders) | 1 | 1
Mitral valve disease mixed (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 21 | 24
Myocardial ischaemia (Cardiac disorders) | 4 | 13
Palpitations (Cardiac disorders) | 2 | 2
Pericardial effusion (Cardiac disorders) | 1 | 2
Pericardial haemorrhage (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 2 | 0
Right ventricular failure (Cardiac disorders) | 0 | 2
Sinoatrial block (Cardiac disorders) | 2 | 0
Sinus arrest (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 2
Sinus node dysfunction (Cardiac disorders) | 6 | 10
Supraventricular extrasystoles (Cardiac disorders) | 1 | 1
Supraventricular tachyarrhythmia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 2
Tachyarrhythmia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Tachycardia induced cardiomyopathy (Cardiac disorders) | 1 | 0
Tricuspid valve disease (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 2 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Cancer gene carrier (Congenital, familial and genetic disorders) | 0 | 1
Congenital ureteric anomaly (Congenital, familial and genetic disorders) | 1 | 0
Corneal dystrophy (Congenital, familial and genetic disorders) | 0 | 1
Muscular dystrophy (Congenital, familial and genetic disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 3
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Otosclerosis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 14 | 8
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Vestibular disorder (Ear and labyrinth disorders) | 1 | 1
Adrenal mass (Endocrine disorders) | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 6 | 5
Hyperthyroidism (Endocrine disorders) | 2 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Thyroiditis (Endocrine disorders) | 1 | 0
Toxic nodular goitre (Endocrine disorders) | 1 | 0
Blepharochalasis (Eye disorders) | 1 | 0
Blindness (Eye disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Cataract (Eye disorders) | 17 | 15
Cataract diabetic (Eye disorders) | 1 | 0
Detachment of macular retinal pigment epithelium (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Ectropion (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 3 | 3
Iridocyclitis (Eye disorders) | 1 | 0
Keratopathy (Eye disorders) | 0 | 1
Macular fibrosis (Eye disorders) | 0 | 3
Maculopathy (Eye disorders) | 1 | 0
Open angle glaucoma (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 0 | 3
Retinal haemorrhage (Eye disorders) | 1 | 2
Retinal tear (Eye disorders) | 0 | 1
Retinal vascular thrombosis (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 2 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 4 | 2
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 10 | 8
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0
Acquired oesophageal web (Gastrointestinal disorders) | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Anal prolapse (Gastrointestinal disorders) | 1 | 0
Anal sphincter atony (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Coeliac disease (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 3 | 2
Colitis ischaemic (Gastrointestinal disorders) | 2 | 2
Colitis microscopic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 8 | 6
Crohn's disease (Gastrointestinal disorders) | 0 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 3
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 3 | 3
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 6
Diverticulum oesophageal (Gastrointestinal disorders) | 0 | 1
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 5 | 3
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Femoral hernia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 6 | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 4 | 9
Gastritis erosive (Gastrointestinal disorders) | 1 | 2
Gastroduodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal mucosal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 | 0
Gastrointestinal stenosis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 1 | 2
Hernial eventration (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 2 | 4
Ileus (Gastrointestinal disorders) | 7 | 3
Inguinal hernia (Gastrointestinal disorders) | 14 | 7
Intestinal angina (Gastrointestinal disorders) | 0 | 1
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 4 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 5 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Intestinal strangulation (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 4 | 5
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Malabsorption (Gastrointestinal disorders) | 0 | 1
Mechanical ileus (Gastrointestinal disorders) | 0 | 2
Melaena (Gastrointestinal disorders) | 2 | 2
Mesenteric artery embolism (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 2
Oesophageal polyp (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatic cyst (Gastrointestinal disorders) | 2 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 4
Pancreatitis acute (Gastrointestinal disorders) | 1 | 4
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1
Peritoneal perforation (Gastrointestinal disorders) | 0 | 1
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Rectal polyp (Gastrointestinal disorders) | 2 | 3
Rectal prolapse (Gastrointestinal disorders) | 1 | 4
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 1
Tongue oedema (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 2 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1
Volvulus of small bowel (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2
Adverse drug reaction (General disorders) | 0 | 1
Asthenia (General disorders) | 3 | 4
Chest pain (General disorders) | 9 | 8
Chronic fatigue syndrome (General disorders) | 1 | 0
Death (General disorders) | 16 | 13
Device dislocation (General disorders) | 3 | 5
Device failure (General disorders) | 0 | 1
Device malfunction (General disorders) | 0 | 2
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Foreign body reaction (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 4 | 4
Hernia (General disorders) | 1 | 1
Incarcerated hernia (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Ischaemic ulcer (General disorders) | 0 | 1
Malaise (General disorders) | 2 | 2
Medical device complication (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 2 | 4
Nodule (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 7 | 5
Oedema peripheral (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 0 | 2
Polyp (General disorders) | 1 | 0
Pyrexia (General disorders) | 4 | 5
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 4 | 1
Ulcer haemorrhage (General disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 2
Bile duct stenosis (Hepatobiliary disorders) | 1 | 2
Bile duct stone (Hepatobiliary disorders) | 0 | 4
Biliary cirrhosis primary (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 2 | 5
Cholangitis (Hepatobiliary disorders) | 4 | 1
Cholecystitis (Hepatobiliary disorders) | 6 | 4
Cholecystitis acute (Hepatobiliary disorders) | 4 | 2
Cholelithiasis (Hepatobiliary disorders) | 22 | 30
Gallbladder necrosis (Hepatobiliary disorders) | 1 | 0
Gallbladder oedema (Hepatobiliary disorders) | 0 | 1
Gallbladder polyp (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 1
Autoimmune disorder (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 0 | 1
Appendiceal abscess (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 4 | 5
Appendicitis perforated (Infections and infestations) | 2 | 1
Arthritis bacterial (Infections and infestations) | 1 | 2
Arthritis infective (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 8 | 7
Bronchitis fungal (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 6 | 6
Cellulitis (Infections and infestations) | 3 | 2
Cholecystitis infective (Infections and infestations) | 0 | 3
Chronic sinusitis (Infections and infestations) | 1 | 0
Chronic tonsillitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 6 | 5
Dengue fever (Infections and infestations) | 2 | 1
Device related infection (Infections and infestations) | 2 | 1
Diverticulitis (Infections and infestations) | 11 | 10
Ear infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 0 | 2
Enterocolitis bacterial (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 4 | 9
Gangrene (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 9 | 9
Gastroenteritis viral (Infections and infestations) | 2 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 1
Haemophilus infection (Infections and infestations) | 1 | 0
Helicobacter gastritis (Infections and infestations) | 2 | 0
Hepatic cyst infection (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 2
Infected skin ulcer (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 2 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 2 | 0
Listeriosis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 0 | 3
Lobar pneumonia (Infections and infestations) | 2 | 4
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 6
Lung infection (Infections and infestations) | 3 | 1
Lymph node tuberculosis (Infections and infestations) | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 1 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 1
Onychomycosis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 2 | 2
Otitis media (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 44 | 48
Pneumonia bacterial (Infections and infestations) | 3 | 4
Pneumonia haemophilus (Infections and infestations) | 1 | 1
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 3 | 2
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 1
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 2
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 5 | 3
Pyelonephritis acute (Infections and infestations) | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 2
Salmonellosis (Infections and infestations) | 1 | 2
Salpingitis (Infections and infestations) | 1 | 0
Salpingo-oophoritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 6 | 15
Septic shock (Infections and infestations) | 5 | 5
Sinusitis (Infections and infestations) | 3 | 1
Skin infection (Infections and infestations) | 0 | 1
Small intestine gangrene (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Stenotrophomonas infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Subdural empyema (Infections and infestations) | 0 | 1
Tick-borne viral encephalitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Tuberculosis of peripheral lymph nodes (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 13 | 11
Urosepsis (Infections and infestations) | 6 | 3
Vaginal infection (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 3 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Cataract traumatic (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 7 | 8
Contusion (Injury, poisoning and procedural complications) | 4 | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 3
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 | 1
Eye penetration (Injury, poisoning and procedural complications) | 2 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 9
Fall (Injury, poisoning and procedural complications) | 13 | 16
Femoral neck fracture (Injury, poisoning and procedural complications) | 16 | 15
Femur fracture (Injury, poisoning and procedural complications) | 16 | 12
Fibula fracture (Injury, poisoning and procedural complications) | 14 | 11
Foot fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 1
Graft complication (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 4 | 6
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 13 | 5
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 1
Injury corneal (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 7 | 6
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 2 | 2
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 4 | 3
Meniscus injury (Injury, poisoning and procedural complications) | 5 | 2
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 3 | 1
Patella fracture (Injury, poisoning and procedural complications) | 5 | 5
Perineal injury (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Postoperative hernia (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 2
Pubis fracture (Injury, poisoning and procedural complications) | 3 | 5
Radiation mucositis (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 25 | 22
Rib fracture (Injury, poisoning and procedural complications) | 7 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 3
Scar (Injury, poisoning and procedural complications) | 0 | 2
Shunt malfunction (Injury, poisoning and procedural complications) | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 5 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 8 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 2
Thermal burn (Injury, poisoning and procedural complications) | 2 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 9
Tibia fracture (Injury, poisoning and procedural complications) | 17 | 12
Toxicity to various agents (Injury, poisoning and procedural complications) | 4 | 2
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 | 2
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 9 | 9
Ulnar nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 2 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 1
Antinuclear antibody positive (Investigations) | 0 | 1
Blood pressure increased (Investigations) | 0 | 1
Blood pressure orthostatic (Investigations) | 1 | 0
Carcinoembryonic antigen increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Investigation (Investigations) | 1 | 0
Occult blood positive (Investigations) | 0 | 1
Protein total decreased (Investigations) | 1 | 0
Troponin increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 3 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 3
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 15
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 4
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 10
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone loss (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 2 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 4 | 7
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 12 | 7
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 4 | 5
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Morphoea (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 79 | 99
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 5 | 3
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 3 | 6
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Plica syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 | 4
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 14 | 22
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 4
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 3
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovial disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenosquamous cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 | 14
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 24
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 12
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dermatofibrosarcoma protuberans (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Diffuse large B-cell lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gingival cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 2
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 13
Lung squamous cell carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Malignant neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Muscle neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nodular fasciitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian epithelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Pelvic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 4
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acoustic neuritis (Nervous system disorders) | 0 | 1
Akinesia (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 3
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 3 | 0
Ataxia (Nervous system disorders) | 1 | 1
Carotid artery occlusion (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 2
Carotid artery thrombosis (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 5
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 2
Cerebral artery embolism (Nervous system disorders) | 1 | 0
Cerebral atrophy (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 5 | 2
Cerebral infarction (Nervous system disorders) | 5 | 17
Cerebral ischaemia (Nervous system disorders) | 6 | 6
Cerebral microangiopathy (Nervous system disorders) | 1 | 0
Cerebral thrombosis (Nervous system disorders) | 8 | 8
Cerebrovascular accident (Nervous system disorders) | 22 | 29
Cerebrovascular disorder (Nervous system disorders) | 1 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 1
Cervicogenic headache (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 3 | 1
Coma (Nervous system disorders) | 0 | 2
Cubital tunnel syndrome (Nervous system disorders) | 0 | 2
Dementia (Nervous system disorders) | 2 | 2
Dementia Alzheimer's type (Nervous system disorders) | 2 | 5
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 5
Dysaesthesia (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 2 | 2
Extrapyramidal disorder (Nervous system disorders) | 0 | 2
Facial paresis (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 2
Haemorrhagic stroke (Nervous system disorders) | 3 | 3
Headache (Nervous system disorders) | 4 | 2
Hemiparesis (Nervous system disorders) | 1 | 2
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 11 | 9
Lacunar infarction (Nervous system disorders) | 2 | 1
Loss of consciousness (Nervous system disorders) | 2 | 3
Lumbar radiculopathy (Nervous system disorders) | 2 | 2
Mental impairment (Nervous system disorders) | 1 | 0
Mononeuropathy multiplex (Nervous system disorders) | 1 | 0
Motor dysfunction (Nervous system disorders) | 1 | 1
Motor neurone disease (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 2 | 1
Nervous system disorder (Nervous system disorders) | 1 | 1
Optic neuritis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Parkinsonism (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 2 | 1
Pseudoradicular syndrome (Nervous system disorders) | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1
Radicular syndrome (Nervous system disorders) | 1 | 2
Radiculitis (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 6 | 12
Seizure (Nervous system disorders) | 2 | 0
Senile dementia (Nervous system disorders) | 2 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 2
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 1
Syncope (Nervous system disorders) | 18 | 20
Tarsal tunnel syndrome (Nervous system disorders) | 1 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 21 | 19
Trigeminal neuralgia (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 3 | 1
Vascular dementia (Nervous system disorders) | 1 | 1
Vascular headache (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 3
Aggression (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 2
Confusional state (Psychiatric disorders) | 6 | 2
Depression (Psychiatric disorders) | 11 | 9
Emotional distress (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 2
Mental disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 1
Schizophrenia, paranoid type (Psychiatric disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 6
Bladder disorder (Renal and urinary disorders) | 0 | 2
Bladder irritation (Renal and urinary disorders) | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 6
Calculus bladder (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 2 | 2
Calculus urethral (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 3 | 1
Cystitis interstitial (Renal and urinary disorders) | 0 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Incontinence (Renal and urinary disorders) | 0 | 1
Mixed incontinence (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 3
Nephropathy (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 5
Stress urinary incontinence (Renal and urinary disorders) | 2 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Ureteric stenosis (Renal and urinary disorders) | 2 | 0
Urethral disorder (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urge incontinence (Renal and urinary disorders) | 1 | 0
Urinary bladder polyp (Renal and urinary disorders) | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 4 | 5
Urinary retention (Renal and urinary disorders) | 1 | 3
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Colpocele (Reproductive system and breast disorders) | 2 | 3
Cystocele (Reproductive system and breast disorders) | 11 | 5
Endometrial atrophy (Reproductive system and breast disorders) | 1 | 0
Endometrial metaplasia (Reproductive system and breast disorders) | 1 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 | 0
Genital prolapse (Reproductive system and breast disorders) | 1 | 0
Mammary duct ectasia (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 4 | 3
Rectocele (Reproductive system and breast disorders) | 4 | 5
Uterine cyst (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 1
Uterine polyp (Reproductive system and breast disorders) | 4 | 4
Uterine prolapse (Reproductive system and breast disorders) | 9 | 9
Vaginal cyst (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 5 | 3
Vulval leukoplakia (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 14 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 19 | 13
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Tonsillar cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Activities of daily living impaired (Social circumstances) | 1 | 0
Physical assault (Social circumstances) | 0 | 1
Anticoagulant therapy (Surgical and medical procedures) | 0 | 1
Arthrodesis (Surgical and medical procedures) | 0 | 1
Benign tumour excision (Surgical and medical procedures) | 1 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 | 1
Chemotherapy (Surgical and medical procedures) | 0 | 1
Hip arthroplasty (Surgical and medical procedures) | 0 | 2
Hospitalisation (Surgical and medical procedures) | 0 | 1
Hysterectomy (Surgical and medical procedures) | 0 | 1
Joint arthroplasty (Surgical and medical procedures) | 1 | 2
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Rehabilitation therapy (Surgical and medical procedures) | 0 | 1
Spinal decompression (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1
Urethral operation (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 5
Aortic dissection (Vascular disorders) | 2 | 0
Aortic stenosis (Vascular disorders) | 5 | 8
Arterial disorder (Vascular disorders) | 0 | 2
Arterial haemorrhage (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 5 | 5
Circulatory collapse (Vascular disorders) | 3 | 1
Deep vein thrombosis (Vascular disorders) | 8 | 8
Embolism venous (Vascular disorders) | 1 | 0
Essential hypertension (Vascular disorders) | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Femoral artery occlusion (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 2 | 3
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 18 | 21
Hypertensive crisis (Vascular disorders) | 7 | 3
Hypotension (Vascular disorders) | 0 | 3
Hypovolaemic shock (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 3
Ischaemia (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 3
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 2
Peripheral artery stenosis (Vascular disorders) | 2 | 0
Peripheral embolism (Vascular disorders) | 2 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 3
Peripheral vascular disorder (Vascular disorders) | 2 | 0
Peripheral venous disease (Vascular disorders) | 0 | 1
Phlebolith (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Subclavian artery occlusion (Vascular disorders) | 0 | 1
Temporal arteritis (Vascular disorders) | 2 | 3
Thrombophlebitis (Vascular disorders) | 1 | 2
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 4 | 3
Varicose vein (Vascular disorders) | 5 | 3
Vasculitis (Vascular disorders) | 2 | 1
Vasculitis necrotising (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/ Denosumab 60 mg Q6M (N=2206) | Denosumab/ Denosumab 60 mg Q6M (N=2343)
Anaemia (Blood and lymphatic system disorders) | 141 | 168
Vertigo (Ear and labyrinth disorders) | 138 | 140
Cataract (Eye disorders) | 319 | 317
Constipation (Gastrointestinal disorders) | 141 | 118
Diarrhoea (Gastrointestinal disorders) | 139 | 152
Bronchitis (Infections and infestations) | 206 | 226
Cystitis (Infections and infestations) | 194 | 212
Influenza (Infections and infestations) | 179 | 192
Nasopharyngitis (Infections and infestations) | 372 | 385
Pneumonia (Infections and infestations) | 137 | 167
Upper respiratory tract infection (Infections and infestations) | 139 | 128
Urinary tract infection (Infections and infestations) | 242 | 250
Contusion (Injury, poisoning and procedural complications) | 181 | 176
Fall (Injury, poisoning and procedural complications) | 240 | 268
Hypercholesterolaemia (Metabolism and nutrition disorders) | 215 | 200
Arthralgia (Musculoskeletal and connective tissue disorders) | 527 | 541
Back pain (Musculoskeletal and connective tissue disorders) | 501 | 493
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 197 | 231
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 332 | 355
Pain in extremity (Musculoskeletal and connective tissue disorders) | 264 | 293
Dizziness (Nervous system disorders) | 173 | 163
Headache (Nervous system disorders) | 121 | 103
Sciatica (Nervous system disorders) | 149 | 165
Depression (Psychiatric disorders) | 135 | 143
Cough (Respiratory, thoracic and mediastinal disorders) | 172 | 168
Hypertension (Vascular disorders) | 460 | 498

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.